CLINICAL TRIAL: NCT06275997
Title: Gastric Cancer and Artificial Intelligence: a National-level Project
Brief Title: GAIN Project: Gastric Cancer and Artificial Intelligence
Acronym: GAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAIN
Record Dates: First submitted 2024-02-02; First posted 2024-02-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel/Crossover Study Model; Patients will be randomized 1:1:1:1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parallel arm 1 (No Intervention): patients will undergo standard high-definition and high-quality upper-GI endoscopy for the detection of gastric lesions with histological mapping according to Sydney system
- Parallel arm 2 (Active Comparator): patients will undergo high-definition and high quality upper-GI endoscopy with real-time assistance by real-time artificial intelligence for the detection of early gastric cancer and gastric dysplasia.
  Interventions: Device: Integration of Artificial Intelligence (AI) assistance to screening gastroscopy
- Cross-over arm 1 (control) (Other): patients will undergo two standard high-definition and high-quality upper-GI endoscopies in tandem: the first will be without Artificial Intelligence assistance, and the second with Artificial Intelligence in order to define the miss rate for standard unassisted upper-GI endoscopy.
  Interventions: Device: Integration of Artificial Intelligence (AI) assistance to screening gastroscopy
- Cross-over arm 2 (Active Comparator): patients will undergo two standard high-definition and high-quality upper-GI endoscopies in tandem: the first will be with Artificial Intelligence assistance, and the second without Artificial Intelligence in order to define the decrease of miss rate when assistance by Artificial Intelligence is implemented.
  Interventions: Device: Integration of Artificial Intelligence (AI) assistance to screening gastroscopy

INTERVENTIONS:
Device: Integration of Artificial Intelligence (AI) assistance to screening gastroscopy — Two novel deep learning systems, namely one for endoscopy and one for pathology, will be trained and validated for the diagnosis of gastric atrophy and metaplasia, including extension and severity. Both of the algorithms will be validated against the cases not used for the training phases. Approximately, the partition will be 5 to 1.
  The benefit and harm of AI-assistance for early diagnosis of gastric cancer will be simulated by developing a Markov model on the natural history of gastric cancer from dysplasia to early and advanced cancer, as well as by the impact of a GS on its natural history. This will also simulate the potential effect of lead- and length-time bias. These data will be incorporated in the simulation model in order to include them in the decision-making process on whether AI-assistance for gastric cancer detection should be or not recommended to health systems.
  Arms: Cross-over arm 1 (control); Cross-over arm 2; Parallel arm 2

SUMMARY:
Our GAIN project comprises four core work packages (WPs): WP1. Nation-level randomized controlled trial; WP2. Development of an innovative AI tool; WP3. Novel microsimulation modelling; WP4. Patient inclusion.

The nation-level multi-center tandem randomized controlled trial (WP1) will contribute to a better understanding of how the real-time AI algorithm can reduce miss rate of early gastric cancer and dysplasia during gastroscopy. Moreover, the innovation project will contribute to development of a novel AI tool (WP2) that can stratify the risk of gastric cancer by identifying in vivo precancerous conditions. Furthermore, a microsimulation modelling will allow us to predict how the use of AI can prevent gastric cancer and affect cost and patients' burdens. The assessment of the balance between benefits and harms is quite crucial especially for this type of medical device because the value of innovative tools is sometimes overestimated due to stakeholders' enthusiasm (WP3). Finally, we will take care of patients' perspective throughout the study project by including patient organization in both WP1, 2, and 3 (WP4).

ELIGIBILITY:
Inclusion Criteria:

* All >60 years-old patients undergoing upper-gastrointestinal (GI) endoscopy for selected indications in Italian areas at high-risk of gastric cancer (Lombardia, Emilia Romagna, Veneto, Friuli-Venezia Giulia).

Exclusion Criteria:

* contraindications to upper-GI endoscopy.
* contraindications to biopsy.
* active upper-GI bleeding or urgent upper-GI endoscopy.
* patients with previous upper-GI surgery involving the stomach.
* patients who were not able or refused to give informed written consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6600 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Miss rate reduction | 2025: 12 months enrollment
  change of the miss rate of early gastric cancer and dysplastic lesions at upper-endoscopy when using AI-assistance (tandem).

SECONDARY OUTCOMES:
Change number of Detections | 1 day procedure and follow up for 2 years
  Change in the detection of early gastric cancer and dysplastic lesions at upper-endoscopy when using AI-assistance (parallel).
patient satisfaction | 2025: during the 12 months enrollment
  Assessment of patient acceptability, satisfaction and tolerance, assessed by questionnaire, towards AI technology for both the detection and the characterization of gastric lesions.